CLINICAL TRIAL: NCT04486053
Title: Effect of Hand Dominance on Functional Outcomes in Pediatric Patients With Flexor Tendon Injuries
Brief Title: Long-term Results of Pediatric Flexor Tendon Injuries
Status: Completed | Type: Observational
Sponsor: Marmara University (Other)
Responsible Party: Sponsor
Other Study IDs: 09.2020.443
Record Dates: First submitted 2020-07-22; First posted 2020-07-24 (Actual); Last update posted 2021-03-17 (Actual); Status verified 2020-11

CONDITIONS: Hand Injuries; Flexor Tendon Injury
Keywords: flexor tendons; children; functional outcome; hand injury
MeSH Terms: conditions — Hand Injuries | interventions — Mass Screening

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with flexor tendon injury: Patients between the ages of 6-18 who have applied to orthopedics emergency department due to hand injury and have been operated with flexor tendon injury, for the last 3 years, were retrospectively scanned from hospital record. Eligible patients for the study were informed about the study by telephone and requested to come hospital for further evaluations including sensory, motor and functional assessments.
  Interventions: Other: Screening

INTERVENTIONS:
Other: Screening — The patients who agreed to participate to the study were assessed with a survey which included age, gender, height, weight and hand dominancy questions. Sensory, motor and functional assessments of the bilateral hand were performed.

SUMMARY:
Hand and upper extremity injuries are among the most common causes of admission of children to the emergency department since they are the most frequently injured part of body following head in pediatric and adolescent population. Although upper extremity fractures and contusions are the main reasons of pediatric hand injuries, tendon injuries are not also uncommon. There are limited data in the literature about the long-term results of children with flexor tendon injury. Therefore, the aim of this study was to evaluate the long-term functional outcomes of children with flexor tendon injury.

DETAILED DESCRIPTION:
Hand and upper extremity injuries are among the most common causes of admission of children to the emergency department since they are the most frequently injured part of body following head in pediatric and adolescent population. Although upper extremity fractures and contusions are the main reasons of pediatric hand injuries, tendon injuries are not also uncommon. While extensor tendon injuries have been reported to be most frequent than flexor tendon injuries for all age groups, the ratio of flexor to extensor tendon injuries is higher in pediatric population than adults and in children younger than 10 years old flexor tendon injuries are more common than extensor tendon injuries.Despite some challenges in the treatment of flexor tendon injuries of children, the outcomes have been reported to be better in children than adults since they have better blood supply, more rapid tendon healing and better remodeling ability of scars and adhesions. However, there is still a risk of permanent morbidities such as significant scarring and stiffness which can cause worse functional outcomes.There are limited data in the literature about the long-term results of children with flexor tendon injury. Therefore, the aim of this study was to evaluate the long-term functional outcomes of children with flexor tendon injury.

ELIGIBILITY:
Inclusion Criteria:

* . Patients between the ages of 6-18 who have applied to orthopedics emergency department due to hand injury and have been operated with flexor tendon injury, for the last 3 years

Exclusion Criteria:

* The patients who had history of bilateral hand injury, delayed surgery, accompanying extensor tendon injury and a follow-up less than six months after injury were excluded from the study.

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Patients with flexor tendon injury
Sampling Method: Non-Probability Sample
Enrollment: 44 (Actual)
Dates: Start 2020-05-15 (Actual); Primary Completion 2020-07-15 (Actual); Study Completion 2020-07-15 (Actual)

PRIMARY OUTCOMES:
Jebson Taylor Hand Function test | Day 0
  Jebsen - Taylor Hand Function Test (JTHFT) was performed on both hands for evaluation of the fine and gross motor functions. It is a standard and objective assessment method of hand functions with activities similar to those performed in daily life. The test consists of 7 subtests. During the test, a separate period is kept for each step. The functions of both hands are evaluated by the following operations; writing, card turning, picking up small common objects, simulated feeding, stacking backgammon-checkers, moving large light objects and moving large heavy objects. Score of each subset is time (seconds) to complete the task and total score is calculated by summing of times for each sub-tests
Grip strength | Day 0
  The grip strength measured using a Baseline Hydraulic Hand Dynamometer according to the recommendations of the American Hand Therapists Association.. It was measured with the shoulder in the adduction, elbow 90 * flexion, forearm neutral and wrist 0-30 * dorsiflexion and 0-15 * ulnar deviation while the person was sitting position. The patient was asked to grasp the dynamometer as tightly as he could. For each side, 3 applications were made with an interval of 20 seconds and the average of these measurements was taken
Pinch Strength | Day 0
  Baseline Hydraulic Pinch Gauge was used to measure pinch strength. The measurement was made in the same position as the grip strength measurement. The pinch gauge was placed between the tip of thumb and the tip of the index finger and the patient was asked to squeeze as strongly as he could. For each side, 3 applications were made with an interval of 20 seconds and the average of these measurements was taken
Semmes -Weinstein Monofilament test | Day 0
  Sensory examination was done with Semmes -Weinstein Monofilament test. This evaluation was started with the smallest monofilament and larger filaments were applied respectively, the test was stopped in the smallest monofilament the patient felt, and this value was recorded. Evaluations were made from the distal tips of the 1st and 2nd finger and the palmar surface of the 2nd metacarpophalangeal joint for the median nerve evaluation (monofilament test 1,2,3, respectively), distal tip of the 5th finger, the palmar surface of the 5th metacarpophalangeal joint and hypothenar area (monofilament test 4, 5, 6, respectively) for ulnar nerve evaluation.

CONTACTS AND LOCATIONS:
Overall Officials: Canan Sanal-Toprak, Asst. Prof, Principal Investigator — Marmara University
Locations (1):
- Marmara University School of Medicine Department of Physical Medicine and Rehabilitation, Istanbul, In the USA Or Canada, Please Select..., Turkey (Türkiye)

REFERENCES:
- [Background] Lee A, Colen DL, Fox JP, Chang B, Lin IC. Pediatric Hand and Upper Extremity Injuries Presenting to Emergency Departments in the United States: Epidemiology and Health Care-Associated Costs. Hand (N Y). 2021 Jul;16(4):519-527. doi: 10.1177/1558944719866884. Epub 2019 Aug 23. PMID 31441332
- [Background] Vadivelu R, Dias JJ, Burke FD, Stanton J. Hand injuries in children: a prospective study. J Pediatr Orthop. 2006 Jan-Feb;26(1):29-35. doi: 10.1097/01.bpo.0000189970.37037.59. PMID 16439897
- [Background] Jeon BJ, Lee JI, Roh SY, Kim JS, Lee DC, Lee KJ. Analysis of 344 Hand Injuries in a Pediatric Population. Arch Plast Surg. 2016 Jan;43(1):71-6. doi: 10.5999/aps.2016.43.1.71. Epub 2016 Jan 15. PMID 26848449
- [Background] Kim JS, Sung SJ, Kim YJ, Choi YW. Analysis of Pediatric Tendon Injuries in the Hand in Comparison with Adults. Arch Plast Surg. 2017 Mar;44(2):144-149. doi: 10.5999/aps.2017.44.2.144. Epub 2017 Mar 15. PMID 28352603
- [Background] Vahvanen V, Gripenberg L, Nuutinen P. Flexor tendon injury of the hand in children. A long-term follow-up study of 84 patients. Scand J Plast Reconstr Surg. 1981;15(1):43-8. doi: 10.3109/02844318109103410. PMID 7268311
- [Background] Nietosvaara Y, Lindfors NC, Palmu S, Rautakorpi S, Ristaniemi N. Flexor tendon injuries in pediatric patients. J Hand Surg Am. 2007 Dec;32(10):1549-57. doi: 10.1016/j.jhsa.2007.08.006. PMID 18070643
- [Background] Cooper L, Khor W, Burr N, Sivakumar B. Flexor tendon repairs in children: Outcomes from a specialist tertiary centre. J Plast Reconstr Aesthet Surg. 2015 May;68(5):717-23. doi: 10.1016/j.bjps.2014.12.024. Epub 2014 Dec 24. PMID 25613292